CLINICAL TRIAL: NCT04565080
Title: Clinical Correlates of COVID-19 Pandemic in Patients With Functional Movement Disorder (FMD) and Parkinson's Disease (PD)
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000159; 000159-N
Record Dates: First submitted 2020-09-24; First posted 2020-09-25 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease; Functional Movement Disorders; COVID-19
Keywords: Parkinson's Disease; Functional Movement Disorders; COVID-19; Natural History
MeSH Terms: conditions — Parkinson Disease; Conversion Disorder; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FMD Patients: adult FMD patients who participated in protocol 07-N-0190
- PD Patients: adult PD patients who participated in protocol 01-N-0206

SUMMARY:
The purpose of this study is to investigate the clinical correlates of the effects of the COVID-19 pandemic on patients with Functional movement disorder (FMD) and Parkinson s Disease (PD).

Primary objectives:

To evaluate the change in neurological symptoms domain of the survey between pre and post-COVID 19 in FMD and PD patients.

Secondary objectives:

* To evaluate the change in total score of the survey between pre and post COVID 19 in FMD and PD patients
* To evaluate the change in other symptom domains of the survey between pre and post COVID 19 in FMD and PD patients. Domains include: Mood/Energy, sleep, symptoms of abnormal movements related or unrelated to primary disease, physical health and exercise related change

Exploratory objectives:

* To evaluate whether there is a modifying effect of disease group in the changes in total score or symptom domains
* To evaluate whether there is a relationship between disease severity and changes in total score or symptom domains
* To evaluate whether there is a correlation between changes across symptom domains
* To evaluate whether there is a correlation in raw score across symptom domains within each period

Research Methods:

Data will be solely collected through the use of online instruments via CiSTAR as a designed questionnaire.

Questionnaire items

A questionnaire aimed at determining the effects of the COVID 19 pandemic and subsequent isolation on functional state of patients with FMD and PD.

The questionnaire items include:

Items investigating Mood/Energy before and after COVID 19 out break

Items investigating Sleep habits before and after COVID 19 out break

Items investigating Neurological symptoms before and after COVID 19 out break

Items investigating daily functioning before and after COVID 19 out break

Items investigating Exercise habits before and after COVID 19 out break

No questionnaire items will be actionable , which are items that would identify an imminent risk for participant safety requiring urgent and immediate medical or psychiatric

DETAILED DESCRIPTION:
The purpose of this study is to investigate the clinical correlates of the effects of the COVID-19 pandemic on patients with Functional movement disorder (FMD) and Parkinson s Disease (PD).

Primary objectives:

To evaluate the change in neurological symptoms domain of the survey between pre and post-COVID 19 in FMD and PD patients.

Secondary objectives:

* To evaluate the change in total score of the survey between pre and post COVID 19 in FMD and PD patients
* To evaluate the change in other symptom domains of the survey between pre and post COVID 19 in FMD and PD patients. Domains include: Mood/Energy, sleep, symptoms of abnormal movements related or unrelated to primary disease, physical health and exercise related change

Exploratory objectives:

* To evaluate whether there is a modifying effect of disease group in the changes in total score or symptom domains
* To evaluate whether there is a relationship between disease severity and changes in total score or symptom domains
* To evaluate whether there is a correlation between changes across symptom domains
* To evaluate whether there is a correlation in raw score across symptom domains within each period

Research Methods:

Data will be solely collected through the use of online instruments via CiSTAR as a designed questionnaire.

Questionnaire items

A questionnaire aimed at determining the effects of the COVID 19 pandemic and subsequent isolation on functional state of patients with FMD and PD.

The questionnaire items include:

Items investigating Mood/Energy before and after COVID 19 out break

Items investigating Sleep habits before and after COVID 19 out break

Items investigating Neurological symptoms before and after COVID 19 out break

Items investigating daily functioning before and after COVID 19 out break

Items investigating Exercise habits before and after COVID 19 out break

No questionnaire items will be actionable , which are items that would identify an imminent risk for participant safety requiring urgent and immediate medical or psychiatric

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. (for FMD subjects only) Clinical diagnosis of Functional movement disorder as confirmed by a movement disorders specialist in subjects previously enrolled in protocol 07-N-0190
  2. (for PD subjects only) Clinical diagnosis of Parkinson s Disease as confirmed by a movement disorders specialist in subjects previously enrolled in protocol 01-N-0206.
  3. Able to give informed consent
  4. Male or female, age 18 and above
  5. Have access to the internet in order to fill out the survey
  6. Have enough fluency in English to be able to read the consent form and take the survey in English

EXCLUSION CRITERIA:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients: adults with clinical diagnosis of Parkinson s Disease as confirmed by a movement disorders specialist in patient s previously enrolled in protocol 01-N-0206.FMD patients: adults with clinical diagnosis of Functional movement disorder as confirmed by a movement disorders specialist in patient s previously enrolled in protocol 07-N-0190.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Change in neurological symptoms domain of the survey between pre and post COVID 19 in FMD and PD patients. | December 2021
  Change in neurological symptoms domain of the survey between pre and post COVID 19 in FMD and PD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States